CLINICAL TRIAL: NCT06277401
Title: High-load Resistance Training Compared With Usual Care for Treatment of Painful Knee Joint Hypermobility in Young Adults: A Randomised Controlled Trial (the HIPEr-Knee Study)
Brief Title: Exercise in Patients With Hypermobile Joints and Knee Pain
Acronym: HIPEr-Knee
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Independent Research Fund Denmark (Industry); Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Behnam Liaghat, Assistant Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT_hypermobile_knee
Record Dates: First submitted 2024-02-09; First posted 2024-02-26 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hypermobility, Joint; Hypermobility Syndrome; Knee Discomfort
Keywords: Hypermobility; Knee pain; Treatment; Randomised controlled trial
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The patients will be kept blind to treatment allocation by being provided with minimal information about the content of the two exercise interventions and the study hypotheses; the patients will be informed that the study compares two different exercise protocols that both include safe exercises to reduce knee pain and increase knee function.
  An independent biostatistician blinded to group allocation will perform the primary RCT analysis. To reduce the risk of interpretation bias, blinded results from the analyses (group A compared with group B) will be presented to all authors, who will agree on two alternative written interpretations before the data manager unblinds the randomisation code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Progressive high-load resistance training program performed twice weekly for 12 weeks
  Interventions: Other: High-load strength training for the knee
- Standard care (Active Comparator): The standard care group will receive instructions on a neuromuscular training program with focus on knee stability and function performed at low intensities to be conducted twice weekly for 12 weeks
  Interventions: Other: Neuromuscular training for the knee

INTERVENTIONS:
Other: Neuromuscular training for the knee — The exercise programme includes exercises identified in literature to target muscles around the knee.
  Arms: Standard care
Other: High-load strength training for the knee — The exercise programme includes exercises identified in literature to target muscles around the knee.
  Arms: Intervention

SUMMARY:
Pain associated with knee joint hypermobility is common in the adult population, but evidence on treatment is sparse. This study investigates if high-load resistance training is superior to usual care in improving activity-related pain in young patients (18-45 years) with hypermobile joints and knee pain.

DETAILED DESCRIPTION:
Knee joint hypermobility is common in the adult population. Patients with knee joint hypermobility and knee pain are typically managed with low intensity resistance training and proprioceptive training to reduce knee pain and improve function, but many patients do not respond well to these treatment strategies. High-load resistance training offers additional benefits to low intensity resistance training, including marked increase in muscle cross-sectional area, neural drive, and increased tendon stiffness, all important components of acquiring active knee joint stability during movement tasks and daily life. Therefore, the primary aim of this randomised controlled trial (RCT) is to investigate if high-load resistance training is superior to usual care in reducing activity-related pain in young patients (18-45 years) with hypermobile joints and knee pain.

ELIGIBILITY:
Inclusion criteria

* Persistent knee pain for ≥ 3 months (self-reported)
* Knee pain ≥ 30mm during the last week using a 0-100 mm visual analogue scale (VAS; 0=no pain and 100=worst imaginable pain) (self-reported)
* Generalised joint hypermobility assessed with the Five-Part Hypermobility Questionnaire (positive ≥ 2/5) (self-reported)
* Local knee joint hypermobility using the passive hyperextension of the knee in standing (positive > 10 degrees of hyperextension) and confirmed in supine lying (heel resting on 20 cm high block on the bench surface), with passive knee hyperextension (positive > 10 degrees) (objectively measured)

Exclusion criteria

* Diagnosed with patellar tendinopathy
* Pregnancy or childbirth within the past year (due to increased levels of relaxin that could affect joint stability)
* Knee surgery within the past year
* Participation in regular structured resistance training within the past six months
* Inability to speak and understand Danish.
* All types of Ehlers-Danlos syndrome
* Other heritable connective tissue disorders such as Marfan syndrome, osteogenesis imperfecta, Loeys-Dietz syndrome, Stickler syndrome, skeletal dysplasias
* Autoimmune rheumatic connective tissue disorders such as lupus, rheumatoid arthritis; Chromosomal conditions such as Fragile X syndrome, Kabuki syndrome, Down syndrome
* Neuromuscular disorders that can cause joints to become unstable, such as multiple sclerosis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale Nominated Activity | Baseline, 6 weeks, 12 weeks (primary endpoint), 12 months
  The primary outcome is the Self-reported knee pain during an activity nominated by patients to be the most aggravating for their present knee pain (VAS nominated activity - VASNA, 0-100, 100 = worse).
  The primary endpoint is at 12-week follow-up.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 12 weeks, 12 months
  Knee injury and Osteoarthritis Outcome Score is a validated knee-specific questionnaire used to assess patient-reported outcomes in the continuum from knee injury to osteoarthritis and is widely used for different types of knee pathology. (0-100, 100 = best)
Adverse events | Up to 12 months
  Adverse events will be defined as any unintended, negative findings, symptom, or illnesses that occur during the study assessments or interventions, whether attributable to the project or not.
Dynamic knee strength | Baseline, 12 weeks
  Dynamic leg strength will be established by a 5-repetition maximum leg press (single leg) by a standardised protocol.
Knee reposition sense | Baseline, 12 weeks
  Sitting active knee joint reposition (proprioception) test will be performed using a HALO Digital Goniometer, to assess mean absolute angle error (AAE)
Single-Leg-Hop for Distance | Baseline, 12 weeks
  The patients will be instructed to hop forward as far as possible and land steadily and stand still for at least three seconds.

OTHER OUTCOMES:
Knee pain past week | Baseline, 6 weeks, 12 weeks, 12 months
  Knee pain for the past week is measured using the Visual Analogue Scale (0-100, 100 = worse)
Tampa scale of Kinesiophobia (TSK) 11 item | Baseline, 12 weeks, 12 months
  Tampa scale of Kinesiophobia is used to measure impression of change in fear of movement from baseline to 16 weeks follow-up. It consists of an 11-item scale where each question is scored on a 4 point Likert scale, with 1 indicating, "strongly disagree" and 4 indicating, "strongly agree". The total scores range from 11-44, with higher scores representing increased fear of movement.
EQ-5D-5L | Baseline, 12 weeks, 12 months
  the European Quality of life-5 Dimensions-5-Level measures change in health related quality of life and includes the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ-5D descriptive system comprises five dimensions (mobility, Self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension is rated using a five-level ordinal scale from no problems to extreme problems. It results in a preference based index that range from states worse than death (<0), to 1 (full health), anchoring dead at 0. A score of one indicates that the participants perceived their health at the best possible state and a score below null that the participants perceived their health worse than death.
EQ VAS | Baseline, 12 weeks, 12 months
  the European Quality of life-5 Dimensions-5-Level measures change in health related quality of life and includes the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ VAS measures change in health related quality of life. It includes a visual analogue scale where own health 'today´ is rated on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
Global perceived effect (GPE) | 12 weeks, 12 months
  To measure the patients self-rated impression of improvement at follow-up the GPE will be used related to knee problems. GPE measures self-rated impression of improvement since baseline assessment on a 7-point scale (1 "worse, an important worsening" to 7 "better, an important improvement)
PASS | 12 weeks, 12 months
  Patient Acceptable Symptom State "When you think of your shoulder function, will you consider your current condition as satisfying? By shoulder function, you should take into account your activities of daily living, sport and recreational activities, your pain and other symptoms and your quality of life". Answered by "yes" or "no".
TF | 12 weeks, 12 months
  Treatment Failure Only answered by patients answering "no" to PASS. "Would you consider your current state as being so unsatisfactory that you consider the treatment to have failed?". Answered by "yes" or "no".
Clinical important difference | 12 weeks, 12 months
  American College of Rheumatology response criteria 20% and 50%
Knee instability questions | Baseline, 12 weeks, 12 months
  Within the last month, have you experienced that your knee was unstable or about to give out? To what extent has the experience of your knee feeling unstable or giving out affected your daily activity level within the last month?
Tendon stiffness | Baseline, 12 weeks
  Stiffness of the patellar tendon is assessed based on corresponding values of tendon force and tendon deformation (measured by use of B-mode ultrasonography). Subgroup of patients (n = 30)
Quadriceps rate of torque development (RTD) | Baseline, 12 weeks
  Rate of torque development in the quadriceps muscle. Subgroup of patients (n = 30)
Patella instability | Baseline, 12 weeks
  Moving patellar apprehension test will be used to assess patella instability. Subgroup of patients (n = 30)
Quadriceps maximal voluntary isometric contraction | Baseline, 12 weeks
  Isometric maximal voluntary contraction in the quadriceps muscle. Subgroup of patients (n = 30)

CONTACTS AND LOCATIONS:
Overall Officials: Behnam Liaghat, PhD, Principal Investigator — University of Southern Denmark; Jonas B Thorlund, PhD, Study Director — University of Southern Denmark
Locations (2):
- Denmark (2):
  - Physiotherapy Clinics Region of Southern Denmark, Odense, Fyn
  - University of Southern Denmark, Odense, Fyn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liaghat B, Bojsen-Moller J, Juul-Kristensen B, Henriksen P, Mohammadnejad A, Heiberg BD, Thorlund JB. High-load strength training compared with standard care treatment in young adults with joint hypermobility and knee pain: study protocol for a randomised controlled trial (the HIPEr-Knee study). BMJ Open. 2024 Oct 16;14(10):e090812. doi: 10.1136/bmjopen-2024-090812. PMID 39414294